CLINICAL TRIAL: NCT03585049
Title: Archive of Vaginal Swabs Microscopic Images for the Development of a Rapid Vaginitis Diagnostic Device
Brief Title: Microscopic Images for the Development of a Rapid Vaginitis Diagnostic Device
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Principal Investigator, Meir Medical Center
Other Study IDs: 077-18-COM1
Record Dates: First submitted 2018-06-30; First posted 2018-07-12 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Vaginitis
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vaginal swabs — The protocol includes the secondary use of vaginal swabs that are primarily used for routine diagnostic assessment in a vulvovaginal clinic

SUMMARY:
The study goal is to create an archive of microscopy images of various vulvovaginal inflammation conditions

DETAILED DESCRIPTION:
During the study, the investigators are planning to make a secondary use of vaginal discharge samples that are primarily taken for routine wet mount microscopic diagnostics in a vulvovaginal clinic at the Women's health center, Ramat-Eshkol, Jerusalem.

In order to create an anonymous archive of digital microscopy images, before each swab is disposed of, the investigator will dilute the collected discharge on the swab with 0.5ml Saline into an Eppendorf tube. The diluted discharge will then be applied onto the GynTools LTD VagX tray that is then scanned by a tabletop scanner. At this point the VagX tray will be washed with water, soap and both the swab and tube will be disposed of.

No of participating patients: 1000 Patients age: 18 years and above. Only from patients capable of signing an informed consent.

ELIGIBILITY:
Inclusion Criteria:

Vulvovaginal complaints

Exclusion Criteria:

Younger than 18y or cannot sign an informed consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 18y that go through a routine vulvovaginal assessment at the clinic
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Creation of microscopy image archive | 1 year
  Collecting 1000 images

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam LevSagie, M.D., Principal Investigator — Clalit Healthcare Services
Locations (1):
- Clalit Women's Health Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD will be collected except for consent forms which will not be shared with other researchers.